CLINICAL TRIAL: NCT04753034
Title: A Multicenter, Randomized, Double-blind, Vehicle-Controlled, Phase 2 Study of TER-101 Topical Ointment to Assess Efficacy and Safety in Subjects With Mild to Moderate Atopic
Brief Title: Study of TER-101 Topical Ointment in Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Teres Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TER101-AD-201
Record Dates: First submitted 2021-01-21; First posted 2021-02-12 (Actual); Results first posted 2022-07-19 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2021-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TER-101 (Experimental): BID (twice daily) application
  Interventions: Drug: TER-101
- Vehicle (Placebo Comparator): Vehicle ointment, BID (twice daily) application
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: TER-101 — Active Comparator
  Arms: TER-101
Drug: Vehicle — Placebo Comparator
  Arms: Vehicle

SUMMARY:
This Phase 2 study will assess efficacy, safety, and tolerability of TER-101 ointment and vehicle twice daily for 28 days in adult and adolescent subjects with mild to moderate atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent or adult subject aged 12 - 65 years.
* Overall IGA score of 2 (mild) or 3 (moderate) at baseline on a 5-point IGA

Exclusion Criteria:

* AD with known hypersensitivity to excipients of TER-101 Ointment
* Subjects who are immunocompromised

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-01-18 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Teres Bio site 05, Scottsdale, Arizona
  - Teres Bio Site 04, Encinitas, California
  - Teres Bio Site 12, North Miami Beach, Florida
  - Teres Bio Site 10, Tampa, Florida
  - Teres Bio Site 02, Clarksville, Indiana
  - Teres Bio Site 01, Louisville, Kentucky
  - Teres Bio site 09, Saint Joseph, Missouri
  - Teres Bio Site 08, High Point, North Carolina
  - Teres Bio Site 11, Wilmington, North Carolina
  - Teres Bio Site 03, College Station, Texas
  - Teres Bio Site 06, Pflugerville, Texas
  - Teres Bio Site 07, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TER-101 | Vehicle
Started | 31 | 32
Completed | 29 | 31
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TER-101 | Vehicle | Total
Number analyzed (Participants) | 31 | 32 | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 3 | 10
  Between 18 and 65 years | 24 | 29 | 53
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 21 | 45
  Male | 7 | 11 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 27 | 29 | 56
  Unknown or Not Reported | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 21 | 15 | 36
  Race: Asian | 5 | 2 | 7
  Race: Black or African American | 4 | 13 | 17
  Race: Other | 0 | 1 | 1
  Race: More than one race | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 31 | 32 | 63
EASI [Mean (Standard Deviation); unit: Scores on a scale] | 7.97 (2.424) | 8.47 (3.016) | 8.22 (2.730)
Overall IGA score [Count of Participants; unit: Participants]
  2 - mild | 8 | 7 | 15
  3 - moderate | 23 | 25 | 48
WI-NRS [Mean (Standard Deviation); unit: scores on a scale] | 5.1 (2.14) | 5.5 (2.58) | 5.3 (2.37)
Total body surface area [Mean (Standard Deviation); unit: Percent of body surface area] | 7.2 (3.58) | 7.8 (3.83) | 7.5 (3.69)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in EASI From Baseline at Day 29
Description: EASI = Eczema Area and Severity Index, EASI combines the assessment of the severity of lesions and the the numerical area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for erythema, induration, lichenification, excoriation are multiplied with value of the area affected and with the percentage of the four body areas.
Time Frame: 29 days
Population: All randomized participants who received at least 1 application of the study treatment and had at least 1 post-baseline efficacy assessment. The treatment group as assigned (randomized) was used for analyses.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Arm/Group | TER-101 | Vehicle
Number analyzed (Participants) | 31 | 32
percent change | -47.37 [-67.088 to -27.653] | -42.10 [-61.476 to -22.721]

2. Secondary Outcome: Changes in EASI Over Time
Description: EASI combines the assessment of the severity of lesions and the area affected into a single total score in the range 0 (no disease) to 72 (maximal disease). To calculate the EASI, the sum of the severity rating (0 to 3 with 3 being the most severe) for erythema, induration, lichenification, excoriation are multiplied with the numerical value of the area affected and with the percentage of the four body areas.
Time Frame: 15 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | TER-101 | Vehicle
Number analyzed (Participants) | 31 | 32
percent | -35.96 [-51.842 to -20.081] | -39.24 [-54.739 to -23.742]

3. Secondary Outcome: Change in IGA From Baseline Over Time
Description: IGA = Investigator Global Assessment (Scale 0 - 4) 0 = Clear
  1. = Almost Clear
  2. = Mild
  3. = Moderate
  4. = Severe
Time Frame: 29 Days
Population: as for outcome 1
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | TER-101 | Vehicle
Number analyzed (Participants) | 31 | 32
score on a scale | -0.7 [-3 to 1] | -0.7 [-3 to 0]

4. Secondary Outcome: Changes in Itch Over Time
Description: The WI-NRS asks subjects to report their worst itch (maximal intensity) during the last 24 hours on an 11-point NRS, ranging from 0 = "no itch at all" to 10 = "worst itch you can imagine".
Time Frame: 29 days
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | TER-101 | Vehicle
Number analyzed (Participants) | 31 | 32
score on a scale | -2.0 [-2.92 to -1.14] | -1.2 [-2.00 to -0.32]

5. Secondary Outcome: Tolerability of TER-101 Ointment vs. Vehicle in Subjects With AD
Description: Sum of erythema, itch, and burning at the time of visit compared to baseline measured on a 0 - 3 scale for each component. A score of 0 indicates no erythema, itch or burning. Higher scores indicate worsening tolerability: 1 (mild), 2 (moderate), 3 (severe)
Time Frame: 29 days
Population: All randomized participants who received at least 1 application of the study treatment. The treatment group for analyses was determined by the treatment received. If any TER-101 was applied, the participant was summarized under the TER-101 treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | TER-101 | Vehicle
Number analyzed (Participants) | 31 | 32
Participants
  Baseline Erythema - none | 17 | 15
  Baseline Erythema - mild | 0 | 2
  Baseline Erythema - moderate | 1 | 2
  Baseline Erythema - Severe | 0 | 0
  Day 29 Erythema - none | 15 | 14
  Day 29 Erythema -mild | 2 | 5
  Day 29 Erythema - moderate | 7 | 7
  Day 29 Erythema - severe | 0 | 0
  Burning/Stinging baseline - none | 22 | 26
  Burning/Stinging baseline - mild | 3 | 3
  Burning/Stinging baseline - moderate | 1 | 1
  Burning/Stinging baseline - severe | 0 | 0
  Burning/Stinging D29 - none | 20 | 24
  Burning/Stinging D29 - mild | 0 | 3
  Burning/Stinging D29 - moderate | 1 | 2
  Burning/Stinging D29 - severe | 1 | 0
  Pruritis - Baseline - none | 14 | 18
  Pruritis - Baseline - mild | 6 | 3
  Pruritis - Baseline - moderate | 2 | 2
  Pruritis - Baseline - severe | 1 | 0
  Pruritis - D29 - none | 13 | 15
  Pruritis - D29 - mild | 7 | 3
  Pruritis - D29 - moderate | 6 | 10
  Pruritis - D29 - severe | 0 | 0

ADVERSE EVENTS:
Time Frame: 29 days
Arm/Group | TER-101 | Vehicle
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/32
Other Adverse Events (participants affected / at risk) | 9/31 | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TER-101 (N=31) | Vehicle (N=32)
Kidney infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TER-101 (N=31) | Vehicle (N=32)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Application site pain (General disorders) | 1 | 1
Product intolerance (General disorders) | 1 | 0
Application site inflammation (General disorders) | 0 | 1
Hangover (General disorders) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Bundle branch block right (Cardiac disorders) | 1 | 0
Eye irritation (Eye disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After database lock, Institution/Investigator may publish trial data generated by Investigator at Institution upon the earlier of: (i) publication of primary Multicenter Publication; or (ii) 18 months after the Trial is completed, if a Multicenter Publication is not submitted by Sponsor for publication within such 18 month period; provided Sponsor has opportunity to review proposed publication or disclosure at least 60 days in advance of its submission to a journal, congress, panel, etc.

DOCUMENTS (2):
  • Study Protocol (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT04753034/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT04753034/SAP_001.pdf